CLINICAL TRIAL: NCT00766805
Title: Endoscopic Variceal Ligation Plus Propranolol And Isosorbide Mononitrate Versus Endoscopic Variceal Ligation Alone For Secondary Prophylaxis Of Variceal Bleeding: A Randomized Controlled Trial
Brief Title: Endoscopic Variceal Ligation (EVL)+ Drugs Versus Endoscopic Variceal Ligation (EVL) Alone For Secondary Prophylaxis
Acronym: Secondary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Dr S K Sarin, Department of Gastroenterology, G B Pant Hospital, New Delhi, India
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2008-PHT-01
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2008-10-06 (Estimated); Status verified 2008-10

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Propranolol; Isosorbide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EVL + Drugs (Active Comparator): Patients randomized to the EVL plus drugs therapy received EVL plus beta-blocker (propranolol) and nitrate (ISMN).
  Interventions: Drug: EVL + Propranolol + Isosorbide 5 mononitrate
- EVL alone (Placebo Comparator): Patients assigned to the EVL group underwent variceal band ligation alone till variceal obliteration.
  Interventions: Other: EVL alone

INTERVENTIONS:
Drug: EVL + Propranolol + Isosorbide 5 mononitrate — Treatment was started with propranolol at a dose of 40 mg twice a day. The heart rate and blood pressure were checked after 12 to 24 hours. The dose of propranolol was increased at increments of 20 to 40 mg per day until the patient achieved a heart rate of 55 bpm, or a maximum dose of 320 mg/day was achieved.ISMN was added at a dose of 10 mg twice a day. The dose was escalated at increments of 10-20 mg/day till a maximum dose of 40 mg/day was reached.
  Arms: EVL + Drugs
Other: EVL alone
  Arms: EVL alone

SUMMARY:
Background: Both endoscopic variceal ligation (EVL) and propranolol are valuable methods for secondary prophylaxis of variceal bleeding. Addition of ISMN to propranolol improves the efficacy of drug therapy. It is hypothesized that a combination of EVL and portal pressure reducing drugs should significantly be better than EVL alone.

Patients and Methods: Patients with history of variceal bleed were randomized to EVL plus drugs (propranolol and ISMN) or EVL alone. EVL was repeated every 3-4 weeks until variceal eradication. Propranolol dose was adjusted to reduce the resting heart rate to 55 bpm. Dose of ISMN was 40 mg/d. Primary end points were rebleed or death. Secondary end points included complications of portal hypertension and the development of serious adverse effects to therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to G B Pant Hospital, New Delhi, with history of hematemesis and/or melena and proven to have esophageal varices as the bleeding source on upper GI endoscopy were included in the study.

Exclusion Criteria:

* A history of undergoing endoscopic sclerotherapy (EST), EVL, or cyanoacrylate injection;
* A history of surgery for portal hypertension;
* Coexisting malignancy;
* Severe cardiopulmonary or renal disease;
* A history of severe side-effects or contraindications to beta-blockers like bronchial asthma, uncontrolled diabetes mellitus, heart failure, peripheral vascular disease, prostatic hypertrophy, arterial hypotension (systolic blood pressure < 100 mm Hg), bradycardia (basal heart rate <55 beats per minute), or complete heart block; and
* Refusal to give consent to participate in the trial.

Ages: 8 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2002-10; Primary Completion 2006-12 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Primary end points of the study were bleeding and death. | During the study period

SECONDARY OUTCOMES:
Complications, UGI bleeding due to causes not related to PHT, and adverse effects that required the discontinuation of therapy. | During the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, G B Pant Hospital, New Delhi, National Capital Territory of Delhi, India